# PROACT Statistical Analysis Plan (SAP)

Project Title: Promoting Smoking Cessation in Lung Cancer Screening Through Proactive

Treatment (PROACT)

Date: February 16, 2023

Project Team: Steven Zeliadt, Spencer Hildie, Claire Chen, Nathan Tomlanovich, Scott

Coggeshall, Jaimee Heffner

#### Contents

| 1. | Study Summary and Aims | 2 |
|---|---|---|
| 2. | Data Sources | 3 |
| 3. | Study Population | 3 |
| 4. | Study Time Period | |
| 5. | Sampling and Randomization | 3 |
| 6. | Study Outcome Measures | 4 |
| 7. | Study Covariates | 5 |
| 8. | Statistical Analyses and Description of Main Tables | 6 |
| 9. | Handling of Missing Data | 9 |
| 10. | Project Links | 9 |
| 11. | Shell Tables and Figures | |

#### 1. Study Summary and Aims

Study purpose:

Investigate an intervention designed to help Veterans stop smoking.

Study design:

Parallel two-arm cluster randomized clinical trial.

**Primary Aim**: Conduct a pragmatic randomized trial among smokers participating in lung cancer screening comparing proactive smoking cessation care with unstructured care. We will assess the differences between the two care approaches on 7-day smoking abstinence 12 months after receipt of screening. Assignment of providers to the two care arms will continue until the study is on track to have 540 patients responding (270 responders per arm) to the 12-month survey. Based on our preliminary findings in a pilot study of proactive care, and related trials in other populations of smokers, we hypothesize that smoking abstinence 12 months after screening will be twice as high (18%) in the proactive group compared to expected abstinence rates in the unstructured group (9%).

#### 2. Data Sources

| | | | Analytic variables of |
|---|---|---|---|
| Data Source | Time Period | Description | Interest |
| CDW | Data Collection | Electronic health<br>record for Dept. Of<br>Veteran Affairs | Smoking status and patient characteristics |
| Surveys | Data Collection | Surveys conducted<br>at 3 and 12 months<br>post LCS | Smoking status, quit attempts, and other patient reported outcomes |

### 3. Study Population

Veterans who smoke being screened for lung cancer at the VA Providence or VA New York Harbor.

| Inclusion Criteria | Exclusion Criteria |
|---|---|
| Current smoker Participant in lung cancer screening | <ul> <li>Patients with urgent findings requiring biopsy/immediate attention on the screening CT</li> <li>Patients with a prior diagnosis of lung cancer or who are receiving active therapy for any cancer other than skin cancer</li> <li>Patients previously diagnosed with cognitive impairment, dementia, or severe behavioral disorders</li> <li>Patients who have an indication in chart review of difficulty communicating or participating in telephone counseling sessions</li> </ul> |

### 4. Sampling and Randomization

This is a cluster randomized two-arm parallel group trial. Randomization occurred at the provider-level. Lists of providers referring patients to lung cancer screening at Study Site A & Study Site B were

prepared. Providers at each site were pair-matched on patient volume and then randomized to either the intervention arm or the control arm. Randomization was performed using random numbers generated with the R programming language.

Following randomization, all patients of enrolled providers who attended lung cancer screening and met eligibility criteria were considered enrolled in the study, with treatment arm corresponding to the randomized treatment arm of their provider.

# 5. Study Outcome Measures

| | | | Assessment<br>Timepoint | | |
|---|---|---|---|---|---|
| Measure (Units) | Comments | Data Type | BL | 3M <sup>1</sup> | 12M <sup>1</sup> |
| Primary Outcome (1) | | | <b>-</b> | | |
| Self-reported smoking cessation at 12 months | Constructed from 12-month survey and EMR data | Binary | | | ✓ |
| Secondary Outcomes (3) | | | | | |
| Experience with Telephone Counseling | Survey only | Binary | | <b>✓</b> | |
| Self-efficacy to quit | Survey only | Likert scale<br>(0-10) | | <b>✓</b> | <b>√</b> |
| Motivational<br>Assessment | Survey only | Likert scale<br>(0-10) | | <b>✓</b> | <b>√</b> |
| Perception of susceptibility to harm | Survey only | Summary<br>Score | | <b>✓</b> | |
| <sup>1</sup> Months post-LCS | | | | | |

# 6. Study Covariates

| | | | Assessment<br>Timepoint | | |
|---|---|---|---|---|---|
| Measure (Units) | Comments | Data Type | BL | 3M <sup>1</sup> | 12M <sup>1</sup> |
| Treatment Assignment | Intervention or Control | Binary | <b>√</b> | | |
| Covariates for primary a | | | | | |
| Site | | Binary | | | |
| Additional covariates for | r primary and secondary sensitivity n | nodels (4) | | | |
| Additional variables coll | ected <sup>2</sup> | | | | |
| Gender | Self-report from screening and baseline questionnaires | Binary | <b>✓</b> | | |
| Marital/partner status | Self-report from screening and baseline questionnaires | Categorical | <b>✓</b> | | |
| Age | Self-report from screening and baseline questionnaires | Continuous | <b>✓</b> | | |
| Highest level of education | Self-report from screening and baseline questionnaires | Ordinal | ✓ | | |
| Current employment status | Self-report from screening and baseline questionnaires | Categorical | ✓ | | |
| Service connection | EHR | Binary | <b>✓</b> | | |
| <sup>1</sup> Months post-LCS | . | | | | |

| | | | Assessment<br>Timepoint | | |
|---|---|---|---|---|---|
| Measure (Units) | Comments | Data Type | BL | 3M¹ | 12M <sup>1</sup> |

#### 7. Statistical Analyses and Description of Main Tables

#### Aim 1 statistical analyses

The primary analysis will be an intent-to-treat based comparison of the two intervention arms. The analysis will be performed at the level of the individual. Clustering of patients within providers will be accounted for in the analysis by the inclusion of a random intercept for provider. The primary analysis will be based on the following random intercept logistic regression model

$$logit^{-1}(P(Y_{ij}|Treatment,Site)) = \beta_0 + \alpha_j + \beta_1 Treatment + \beta_2 Site$$

Where  $Y_{ij}$  is an indicator variable for whether the  $i^{th}$  patient of the  $j^{th}$  provider had quit smoking at 12 months, *Treatment* is a binary indicator for assigned treatment arm, and *Site* is a binary indicator for VA medical center (New York Harbor or Providence). The  $\alpha_j$  represent random intercepts for each provider and are assumed to follow a common N(0,  $\sigma^2$ ) distribution. We will report point estimates and 95% confidence intervals for the odds ratio  $\exp(\beta_1)$ . Confidence intervals will be computed using bootstrap methods. A test of the hull hypothesis of no association ( $\beta_1 = 0$ ) will be performed using a likelihood ratio test. A p-value of less than 0.05 will be taken as sufficient evidence to reject the null hypothesis of no association.

Analyses for secondary outcomes will use models with similar predictor terms but with different link functions depending on the outcome. The table below describes model types in more detail for each outcome.

| | | | Independent | Model | Statistical |
|---|---|---|---|---|---|
| Analysis | Description | Outcome | Variable(s) | type | Test |
| | | | Binary | Logistic | |
| | | Indicator of | treatment | regression | |
| | Smoking | smoking | indicator; | with | |
| Primary outcome | cessation at | abstinence | Binary site | random | |
| | 12 months | at 12 | indicator; | intercept | |
| | | months | Categorical | for | |
| | | | provider | provider | |

| Analysis | Description | Outcome | Independent<br>Variable(s) | Model<br>type | Statistical<br>Test |
|---|---|---|---|---|---|
| 7 maryon | Description | - Cuttomic | (clustering variable) | турс | rest |
| Secondary outcome | Use of smoking cessation support within 3 months of LCS | Indicator for receipt of medication or behavioral counseling | Binary<br>treatment<br>indicator;<br>Binary site<br>indicator;<br>Categorical<br>provider<br>(clustering<br>variable) | Logistic<br>regression<br>with<br>random<br>intercept<br>for<br>provider | |
| Secondary outcome | Use of smoking cessation support within 12 months of LCS | Indicator for receipt of medication or behavioral counseling | Binary<br>treatment<br>indicator;<br>Binary site<br>indicator;<br>Categorical<br>provider<br>(clustering<br>variable) | Logistic<br>regression<br>with<br>random<br>intercept<br>for<br>provider | |
| Secondary outcome | Smoked in<br>the last 7<br>days (3<br>month<br>survey) | Indicator for smoking | Binary<br>treatment<br>indicator;<br>Binary site<br>indicator;<br>Categorical<br>provider<br>(clustering<br>variable) | Logistic<br>regression<br>with<br>random<br>intercept<br>for<br>provider | |
| Secondary outcome | Smoked in<br>the last 7<br>days (12<br>month<br>survey) | Indicator for smoking | Binary<br>treatment<br>indicator;<br>Binary site<br>indicator;<br>Categorical<br>provider<br>(clustering<br>variable) | Logistic<br>regression<br>with<br>random<br>intercept<br>for<br>provider | |
| Secondary outcome | Quit<br>attempts<br>since LCS ( 3<br>months) | | | | |
| Secondary outcome | Tried to reduce or cutdown | Indicator for<br>Yes | Binary<br>treatment<br>indicator; | Logistic<br>regression<br>with | |

| | | | Independent | Model | Statistical |
|---|---|---|---|---|---|
| Analysis | Description since LCS ( 3 | Outcome | Variable(s) Binary site | <b>type</b> random | Test |
| | 3 months | | indicator; | intercept | |
| | | | Categorical | for | |
| | | | provider | provider | |
| | | | (clustering | | |
| | Ouit | | variable) | | |
| | Quit attempts | | | | |
| Secondary outcome | since LCS ( 12 | | | | |
| | months) | | | | |
| | | | Binary | | |
| | | | treatment | Logistic | |
| | Tried to | | indicator; | regression | |
| Secondary outcome | reduce or cutdown | Indicator for | Binary site indicator; | with<br>random | |
| Secondary outcome | since LCS ( 12 | Yes | Categorical | intercept | |
| | months | | provider | for | |
| | | | (clustering | provider | |
| | | | variable) | | |
| | | Ordered | Binary | Ordered | |
| | | categorical | treatment | logistic | |
| | | (A little/not at all | indicator;<br>Binary site | regression | |
| Secondary outcome | Support | satisfied, | indicator; | with | |
| Secondary successive | Satisfaction | somewhat | Categorical | random | |
| | | satisfied, | provider | intercept<br>for | |
| | | very | (clustering | provider | |
| | | satisfied) | variable) | provider | |
| | | | Binary<br>treatment | Linear | |
| | | | indicator; | regression | |
| | | Score on | Binary site | with | |
| Secondary outcome | Motivation to | motivation | indicator; | random | |
| | quit | to quit scale | Categorical | intercept | |
| | | | provider | for | |
| | | | (clustering | provider | |
| | | | variable) | Linear | |
| | | | Binary<br>treatment | regression | |
| | C 10 00 | Score on | indicator; | with | |
| Secondary outcome | Self-efficacy | self-efficacy | Binary site | random | |
| | for quitting | scale | indicator; | intercept | |
| | | | Categorical | for | |
| | | | provider | provider | |

| | | | Independent | Model | Statistical |
|---|---|---|---|---|---|
| Analysis | Description | Outcome | Variable(s) | type | Test |
| | | | (clustering | | |
| | | | variable) | | |
| | | | Binary | | |
| | | Score on susceptibility scale | treatment | Linear | |
| | Perceived<br>susceptibility<br>to lung<br>cancer | | indicator; | regression | |
| | | | Binary site | with | |
| Secondary outcome | | | indicator; | random | |
| | | | Categorical | intercept | |
| | | | provider | for | |
| | | | (clustering | provider | |
| | | | variable) | | |

### 8. Handling of Missing Data

In descriptive statistics, we will describe the extent of missing data. We will examine whether there is differential missingness in outcomes across treatment arms and sites. We will assess the extent to which the distributions of patient characteristics differ between those with the primary outcome and those without the primary outcome.

Patients may have missing data due to survey non-response or missing EHR data. The primary analysis will be a complete-case analysis among those who have a smoking status at 12 months. In sensitivity analyses, we will adapt a method to examine the impact of non-ignorable missingness on the study's primary conclusions. We will use the following model, which incorporates a Missing Not at Random (MNAR) missingness mechanism through a sensitivity parameter representing the odds ratio of smoking cessation between people with missing outcomes and people without missing outcomes.

$$logit^{-1}(P(Smoking)) = \beta_0 + \beta_1 Tx + \beta_2 Site + \beta_3 Missing$$

### 9. Project Links

Clinical Trials Website:

https://clinicaltrials.gov/ct2/show/NCT03612804